CLINICAL TRIAL: NCT01624636
Title: A Multiple Dose, Two-cohort Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Intravenous LFG316 in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Safety and Tolerability of Intravenous LFG316 in Wet Age-related Macular Degeneration (AMD).
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLFG316A2201
Record Dates: First submitted 2012-05-03; First posted 2012-06-21 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-03

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: AMD; Age-related Macular Degeneration; Wet AMD; Neovascular AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- LFG316: 10 mg/kg (2 doses in cohort 1) (Experimental)
  Interventions: Drug: LFG316
- LFG316: 20 mg/kg (2 doses in cohort 1, 3 doses in cohort 2). (Experimental)
  Interventions: Drug: LFG316

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: LFG316
  Arms: LFG316: 10 mg/kg (2 doses in cohort 1)
Drug: LFG316
  Arms: LFG316: 20 mg/kg (2 doses in cohort 1, 3 doses in cohort 2).

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of successive intravenous (IV) doses of LFG316 in eligible patients with neovascular age-related macular degeneration (AMD)

ELIGIBILITY:
Inclusion Criteria:

- Active choroidal neovascular AMD in at least one eye.

Exclusion Criteria:

* Retinal disease other than AMD that, in the investigator's opinion, would interfere with safety or study conduct.
* Choroidal neovascularization due to a cause other than AMD.
* In the study eye, media opacity that, in the investigator's opinion, would interfere with study conduct.
* Any disease or concomitant (or recent) medication expected to cause systemic immunosuppression.
* History of meningococcal meningitis in the past 10 years, or any history of recurrent meningitis.
* History of hospitalization for pneumococcal pneumonia within the past 3 years.
* History of serious systemic infection within the past 12 months.
* Any of the following treatments to the study eye within 7 days prior to study drug dosing: ranibizumab (Lucentis), bevacizumab (Avastin), pegaptanib (Macugen), or other VEGF inhibitor.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of anti-vascular endothelial growth factor (anti-VEGF) retreatment vs time | Day 1 to Day 113 (starting from the day of dosing until the end of the study)
  Number of retreatments with anti-VEGF treatments will be recorded.
Number and percentage of patients with adverse events. | Day 1 to Day 113 (starting from the day of dosing until the end of the study)
  Adverse events will be determined based on descriptive analyses of vital signs, ECG evaluation, and clinical safety laboratory evaluations. All abnormalities will be flagged and summary statistics will be provided by treatment and visit/time.Will be tabulated by body system and preferred term with a breakdown by treatment.

SECONDARY OUTCOMES:
Effect of LFG316 on visual acuity | Day 1 to Day 113
  "Early Treatment Diabetic Retinopathy Study" (ETDRS best corrected visual acuity measured under ETDRS conditions). Number of letters correctly read will be recorded.
Effect of LFG316 on central retinal thickness, choroidal neovascular membrane area and drusen volume. | Day 1 to Day 113
  summary statistics will be provided by treatment group, cohort and visit/time. Treatment effect will be assessed by comparison of mean change from baseline to Day 85 of patients who received or did not receive anti-VEGF therapy.
Serum concentrations of total LFG316 versus time | Days 1, 8, 15, 22, 29, 43, 57, 78, 85 and 113 for both cohorts.
  Blood samples will be collected.
Serum concentration of pharmacodynamic parameters (Weislab and C5) versus time | screening and Days 1, 8, 15, 22, 29, 43, 57, 78, 85 and 113 (for both cohorts).
  Blood samples will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Winter Haven, Florida
  - Novartis Investigative Site, Cleveland, Ohio

REFERENCES:
- See also: Results for CLFG316A2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=11763